CLINICAL TRIAL: NCT03658538
Title: Motivational Interviewing and Air Cleaners for Smokers With COPD (MOVE COPD)
Acronym: MOVE-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB00185955; R01ES029512 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: COPD, Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Treatment (Active Comparator): The active treatment arm will receive two portable active HEPA air cleaners as well as 4 sessions of phone based motivational interviewing to support a home smoking ban and SHS reduction (in addition to the smoking cessation counseling received by all study participants).
  Interventions: Device: Active HEPA Air Cleaner; Behavioral: Motivational interviewing
- Control Arm (Sham Comparator): Homes in the control group will receive Sham air cleaners that have the internal HEPA filter removed, but which will run normally, including similar noise, airflow and overall appearance compared to active air cleaners, thus blinding participants to filter status. The control arm will not receive phone based motivational interviewing to support a home smoking ban and SHS reduction, they will receive only smoking cessation counseling.
  Interventions: Device: Sham Air Cleaner

INTERVENTIONS:
Device: Active HEPA Air Cleaner — The active treatment arm will receive two active air cleaners with HEPA and carbon filters to support a home smoking ban and SHS reduction.
  Arms: Active Treatment
Behavioral: Motivational interviewing — The active treatment arm will receive 4 sessions of phone based motivational interviewing to support a home smoking ban and SHS reduction (in addition to the smoking cessation counseling received by all study participants).
  The Control arm will receive only continued counseling for smoking cessation.
  Arms: Active Treatment
Device: Sham Air Cleaner — The Control arm will receive sham air cleaners
  Arms: Control Arm

SUMMARY:
COPD is characterized by lung injury and inflammation caused by noxious particles and gases, including those emanating from cigarette smoke and air pollution. Despite the clear detrimental impact of poor air quality on respiratory outcomes, regardless of smoking status, to investigators' knowledge, there are no studied environmental interventions targeting indoor air quality to improve respiratory health of smokers, thus ignoring a potential target for harm reduction. Investigators propose a randomized controlled intervention trial to test whether targeted reductions of multiple indoor pollutants (PM, SHS and NO2) in homes of smokers with COPD will improve respiratory outcomes. Investigators have chosen a potent, multimodal intervention (active air cleaners + Motivational intervention for SHS reduction) in order to maximize the opportunity to prove that there is a health benefit to active smokers with COPD from indoor air pollution reduction.

DETAILED DESCRIPTION:
People with COPD who have higher exposure to indoor pollutants, including particulate matter (PM), second hand smoke (SHS), and nitrogen dioxide (NO2) have worse respiratory morbidity including a higher risk of exacerbations. These effects are not obscured by smoking habit. Unfortunately, despite the clear detrimental impact of poor air quality on respiratory outcomes, regardless of smoking status, to investigators' knowledge, there are no studied environmental interventions targeting indoor air quality to improve respiratory health of smokers, thus ignoring a potential target for harm reduction.

Investigators propose a randomized controlled intervention trial to test whether targeted reductions of multiple indoor pollutants (PM, SHS and NO2) in homes of smokers with COPD will improve respiratory outcomes. Investigators have chosen a potent, multimodal intervention in order to maximize the opportunity to prove that there is a health benefit to active smokers with COPD from indoor air pollution reduction. After a one-month run in period in which all participants will receive smoking cessation strategies including Motivational Interviewing (MI) and nicotine replacement therapy, participants unable to quit smoking (n=120) will have 1:1 randomization to receive either 1) multi-component environmental intervention (active "high-efficiency particulate air"(HEPA) air cleaners + MI intervention for SHS reduction) or 2) sham air cleaners. Referrals to community resources for additional support will also be provided. Investigators aim to determine whether a multi-component environmental intervention (targeting PM, SHS and NO2 reduction) will improve respiratory morbidity (i.e., symptoms, quality of life, lung function and exacerbation risk) (Specific Aim #1) and intermediate outcome measures (i.e., markers of airway and systemic inflammation and oxidative stress) (Specific Aim #2) in smokers with COPD. Investigators anticipate that results from this study will inform clinical practice guidelines and health care policies aimed at reducing COPD morbidity and may have broader implications for indoor environmental recommendations for smokers with chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years,
* Physician diagnosis of COPD,
* Global Initiative for Obstructive Lung Disease (GOLD) Stage II-IV disease with Forced Expiratory Volume (FEV1)/ Forced Vital Capacity (FVC) <70% and FEV1 (% predicted) <80%. IF FEV1/FVC <70% and FEV1 (% predicted) ≥ 80%, additional requirement will apply/will be asked: COPD Assessment Test (CAT) score ≥ 10 OR exacerbation history during the last 12 months.
* Tobacco exposure ≥ 10 pack-years
* Current smoker with an exhaled Carbon Monoxide (eCO) ≥ 7 ppm to confirm smoking status. We will employ a combination of self-report and a biochemical marker to identify former-smokers. (If no eCO performed due to COronaVIrus Disease-19 (COVID-19) pandemic safety reasons, we will rely on self-report smoking status and self-report 7-day abstinence questionnaire answers)
* No home smoking ban. IF smoking is not allowed indoor (inside participant's home) then a "home air quality assessment visit" may be done.

Exclusion Criteria:

* Chronic systemic corticosteroids,
* Other chronic lung disease including asthma,
* Living in location other than home (e.g., long term care facility)
* Home owner or occupant planning to move or change residence within study period.
* Air Cleaners drop off (home visits temporary criteria due to COVID-19).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N Hansel, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the Baltimore/Washington are (MD, USA) between June 2019 and January 2024.
Pre-assignment Details: Of the 144 enrolled participants, 121 met inclusion criteria. 1 of those participants dropped out prior to completing the baseline visit and was excluded from analysis.
Groups:
- Active Treatment: The active treatment arm will receive two portable active High-Efficiency Particulate Air (HEPA) air cleaners as well as 4 sessions of phone based motivational interviewing to support a home smoking ban and secondhand smoking (SHS) reduction in addition to the smoking cessation counseling received by all study participants.
  Active HEPA (high-efficiency particulate air) Air Cleaner: The active treatment arm will receive two active air cleaners with HEPA (high-efficiency particulate air) and carbon filters to support a home smoking ban and SHS (secondhand smoking) reduction.
  Motivational interviewing: The active treatment arm will receive 4 sessions of phone based motivational interviewing to support a home smoking ban and SHS (secondhand smoking) reduction (in addition to the smoking cessation counseling received by all study participants).
  The Control arm will receive only continued counseling for smoking cessation.
- Control Arm: Homes in the control group will receive Sham air cleaners that have the internal high-efficiency particulate air (HEPA) filter removed, but which will run normally, including similar noise, airflow and overall appearance compared to active air cleaners, thus blinding participants to filter status. The control arm will not receive phone based motivational interviewing to support a home smoking ban and secondhand smoking (SHS) reduction, they will receive only smoking cessation counseling.
  Sham Air Cleaner: The Control arm will receive sham air cleaners
Period: Overall Study
Arm/Group | Active Treatment | Control Arm
Started | 59 | 61
Completed | 48 | 51
Not Completed | 11 | 10
Not completed — Death | 2 | 1
Not completed — Cancer diagnosis | 1 | 0
Not completed — Change residence | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Unblinded | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Incomplete clinical visit at 6 months due to illness | 1 | 0
Not completed — Evicted from home | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: The active treatment arm will receive two portable active HEPA air cleaners as well as 4 sessions of phone based motivational interviewing to support a home smoking ban and SHS reduction (in addition to the smoking cessation counseling received by all study participants).
  Active HEPA Air Cleaner: The active treatment arm will receive two active air cleaners with HEPA and carbon filters to support a home smoking ban and SHS reduction.
  Motivational interviewing: The active treatment arm will receive 4 sessions of phone based motivational interviewing to support a home smoking ban and SHS reduction (in addition to the smoking cessation counseling received by all study participants).
  The Control arm will receive only continued counseling for smoking cessation.
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Control Arm | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.59 (8.0) | 62.18 (6.0) | 62.88 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 75
  Male | 24 | 21 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 40 | 74
  White | 20 | 21 | 41
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Some College Education or Above [Count of Participants; unit: Participants] | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life -St. George's Respiratory Questionnaire (SGRQ)
Description: St. George's Respiratory Questionnaire (SGRQ). The total score is from 0 to 100. Higher scores indicate more quality of life limitations.
Time Frame: Baseline and 6 months
Population: The difference in the overall number of participants analyzed is due to participants not having SGRQ data collected in either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 47 | 51
score on a scale | -2.9 [-5.6 to -0.2] | 1.5 [-1.1 to 4.1]
Statistical Analysis 1: Comparison: Active Treatment vs Control Arm; Test type: Superiority; p = 0.025, Generalized Linear Mixed Model (GLMM) — P-value corresponds to the statistical significance of the group difference (active vs. control) in the primary outcome, and was not adjusted for the multiple comparison and based on the a priori threshold for statistical significance (P<0.05); The analysis was adjusted for covariates; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-8.2 to -0.5]

2. Primary Outcome: Change in Dyspnea as Assessed by the University of California San Diego Shortness of Breath Questionnaire (SDSOBQ)
Description: Dyspnea will be assessed using the University of California San Diego Shortness of Breath Questionnaire (SDSOBQ). The SDSOBQ scoring will range from 0 to 120 (with higher scores indicating greater difficulty breathing).
Time Frame: Baseline and 6 months
Population: The difference in the overall number of participants analyzed is due to participants not having the University of California San Diego Shortness of Breath Questionnaire (SDSOBQ) data collected n either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 48 | 51
score on a scale | -4.8 [-9.3 to -0.3] | 1.3 [-3.0 to 5.7]
Statistical Analysis 1: Comparison: Active Treatment vs Control Arm; Test type: Superiority; p = 0.061, Generalized Linear Mixed Model (GLMM) — [p-value comment as in outcome 1, analysis 1]; The analysis was adjusted for covariates

3. Secondary Outcome: Change in COPD Health Status Will be Assessed by the COPD Assessment Test (CAT)
Description: Change in COPD health status will be assessed by the COPD assessment test (CAT). The total score is from 0 to 40. Higher scores indicate worse COPD control.
Time Frame: Baseline and 6 months
Population: The difference in the overall number of participants analyzed is due to participants not having the COPD assessment test (CAT) data collected in either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 48 | 51
score on a scale | -1.8 [-3.2 to -0.4] | 1.0 [-0.3 to 2.4]

4. Secondary Outcome: Change in Dyspnea (Breathlessness) as Assessed by the Modified Medical Research Council Questionnaire (mMRC)
Description: Dyspnea (breathlessness) assessed by the modified Medical Research Council questionnaire (mMRC). Mean Score range is 0-4. Higher scores indicate worse COPD control.
Time Frame: Change from baseline and 6 months post-randomization
Population: The difference in the overall number of participants analyzed is due to participants not having the modified Medical Research Council questionnaire (mMRC) data collected in either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 48 | 51
score on a scale | -0.3 [-0.6 to -0.03] | 0.1 [-0.1 to 0.4]

5. Secondary Outcome: Difference in the Proportion (Probability) of Health Care Utilization Due to COPD-related Exacerbations
Description: Questionnaire administered to collect participant's self report of Health Care Utilization (HCU) episodes due to COPD-related exacerbation (including need for oral corticosteroids or antibiotics for worsening respiratory symptoms, emergency department (ED) visit or hospitalization). This questionnaire will be administered at baseline and during the 6 months of follow-up. The HCU number could range from 0 (zero/no episode reported) to 1 (1 or more episodes reported) during the 6 months follow-up.
Time Frame: From Baseline to 6 months
Population: The difference in the overall number of participants analyzed is due to participants not completing (data not collected) the exacerbation survey between baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: Proportion of events
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 53 | 51
Proportion of events
  Severe Exacerbations | 0.11 [0.03 to 0.18] | 0.09 [0.01 to 0.16]
  Moderate Exacerbations | 0.07 [0.004 to 0.14] | 0.19 [0.08 to 0.29]

6. Secondary Outcome: Lung Function as Assessed by the Post Forced Expiratory Volume in 1 Second (FEV1%) Predicted
Description: Pulmonary function testing will be assessed as FEV1% predicted, that is FEV1, adjusted for age, height, race and sex
Time Frame: Baseline and 6 months
Population: The difference in the overall number of participants analyzed is due to participants not having FEV1 data collected in either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: FEV1 percent predicted
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 38 | 45
FEV1 percent predicted | -1.2 [-3.7 to 1.2] | -0.8 [-3.0 to 1.4]

7. Secondary Outcome: Change in the Clinical COPD Questionnaire (CCQ)
Description: The Clinical COPD Questionnaire (CCQ) will be administered to evaluate health status in patients with COPD. The CCQ is a 10-item questionnaire, health-related quality of life questionnaire (HRQoL) with good psychometric properties. The total score ranges from 0 to 6, where a higher scores indicates a worse health status.
Time Frame: Baseline and 6 months
Population: The difference in the overall number of participants analyzed is due to participants not having the Clinical COPD Questionnaire (CCQ) data collected in either baseline and/or 6 months period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Treatment | Control Arm
Number analyzed (Participants) | 47 | 51
score on a scale | -0.2 [-0.5 to -0.003] | -0.8 [-3.0 to 1.4]

8. Other Pre Specified Outcome: Change in Systemic Markers of Inflammation in Serum (Interleukin-8)
Description: Change in systemic markers of inflammation in serum (Interleukin-8) will be measured by Interleukin-8 concentration in serum (units/mg).
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Systemic Markers of Inflammation in Serum (C-reactive Protein)
Description: Change in Systemic markers of inflammation in serum (C-reactive protein) will be measured by C-reactive protein concentration in serum and it will be expressed in: mg/l
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Markers of Oxidative Stress in Urine (8-isoprostane)
Description: Change in Markers of oxidative stress in urine (8-isoprostane) will be measured by 8-isoprostane concentration in urine (pg/ml).
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From randomization up to 6 months
Arm/Group | Active Treatment | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/59 | 1/61
Serious Adverse Events (participants affected / at risk) | 4/59 | 3/61
Other Adverse Events (participants affected / at risk) | 3/59 | 1/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=59) | Control Arm (N=61)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Gastric Mass (Gastrointestinal disorders) | 1 | 0
Syncope (Hypotension and dehydration) (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Influenza (Hospitalized) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Knee Scope Surgery (Surgical and medical procedures) | 0 | 1
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=59) | Control Arm (N=61)
Hypertension (Elevated high blood pressure) (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Adverse Reaction (Palpitations/jitters) to the Nicotine Replacement Therapy (Gum) (Injury, poisoning and procedural complications) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03658538/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03658538/SAP_001.pdf